CLINICAL TRIAL: NCT07103304
Title: Liquid Biopsies for Detecting Somatic Mutations in Sporadic Cerebral Arteriovenous Malformations. Contribution of Sampling From the Drainage Vein of the Malformation.
Brief Title: Liquid Biopsies for Detecting Somatic Mutations in Sporadic Cerebral Arteriovenous Malformations.
Acronym: BioMAV2
Status: Not yet recruiting | Type: Observational
Sponsor: University Hospital, Rouen (Other)
Responsible Party: Sponsor
Other Study IDs: 2023/0310/OB; N° IDRCB : 2025-A00757-42 (Other: ANSM)
Record Dates: First submitted 2025-07-23; First posted 2025-08-05 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-06

CONDITIONS: Cerebral Arteriovenous Malformations
Keywords: embolisation; Search for activating somatic genetic mutations
MeSH Terms: conditions — Intracranial Arteriovenous Malformations

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Biospecimen Retention: Samples With DNA — Whole blood drawn from a peripheral vein at the start and end of embolisation via the venous catheter used by the anaesthesia team as part of routine care for Research into somatic genetic mutations that activate the RAS/RAF/MEK/ERK (MAPK) signalling pathway in cAVMs
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Search for activating somatic genetic mutations — This research aims to evaluate the genetic mutations identified by liquid biopsies on the drainage vein of AVMs, and the prevalence of each mutation.
  These liquid biopsies will be performed during the embolisation procedure by sampling the drainage vein of the malformation and peripheral venous blood (no additional procedures compared to standard care).

SUMMARY:
Cerebral arteriovenous malformations (CAVMs) are abnormal vessels located on the surface of the brain or within the cerebral parenchyma, causing abnormal communication between the arterial and venous networks, without the interposition of the capillary bed. The main risk associated with these malformations is rupture, which causes intracranial bleeding and can lead to serious sequelae or even death. CAVMs (except those of clearly identified genetic origin [< 5%], such as mutations associated with Rendu-Osler disease) have long been considered to be of non-genetic origin.

However, somatic genetic mutations that activate the RAS/RAF/MEK/ERK (MAPK) signalling pathway have recently been identified in surgical specimens of cAVMs. Furthermore, targeted inhibition of this pathway is effective in treating these malformations in animals and appears to be effective in extracranial arteriovenous malformations, particularly superficial ones.

DETAILED DESCRIPTION:
Next-generation sequencing of circulating DNA in liquid biopsies is a promising new and minimally invasive approach for studying the presence of mutations in arteriovenous malformations.

The goal of treating a cAVM is to obliterate the malformation in order to prevent or avoid the risk of haemorrhage. Several therapeutic modalities may be used, which can be combined: microsurgery, endovascular embolisation, and/or radiosurgery. However, these are invasive treatments that are not without risk.

The detection of mutations by liquid biopsies would enable the development of targeted, non-invasive drug therapies against these cAVMs.

The population consists of patients aged 18 years or older with cAVMs, for whom treatment by venous embolisation was recommended during a multidisciplinary consultation meeting.

This research focuses on identifying somatic genetic mutations that activate the RAS/RAF/MEK/ERK (MAPK) signalling pathway in cAVMs. These mutations have already been identified in surgical specimens. This research aims to evaluate the genetic mutations identified by liquid biopsies on the drainage vein of cAVMs and the prevalence of each mutation.

These liquid biopsies will be performed during embolisation surgery by sampling the drainage vein of the malformation and peripheral venous blood (no additional procedures compared to usual care).

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Treated for cAVM
* Indication for embolisation treatment decided upon during a multidisciplinary team meeting (MDT)
* Venous embolisation, with or without arterial embolisation
* Patients informed about the study and willing to participate

Exclusion Criteria:

* Extra-cerebral arteriovenous malformations
* Under legal protection measures (guardianship/curatorship, etc.)
* Pregnancy
* Not eligible for intravenous treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The population consists of patients aged 18 years or older with cAVMs, for whom treatment by venous embolisation was recommended during a multidisciplinary consultation meeting.
Sampling Method: Probability Sample
Enrollment: 16 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2028-01-02 (Estimated); Study Completion 2028-04-01 (Estimated)

PRIMARY OUTCOMES:
Evaluate genetic mutations identified by liquid biopsies on the drainage vein of AVMs. | Embolisation procedure (D0), i.e. a maximum of 45 days after the patient has agreed to participate
  determination of each mutation identified in the drainage vein of AVMs,
Assessment of the prevalence of each mutation identified by liquid biopsies on the drainage vein of AVMs | Embolisation procedure (D0), i.e. a maximum of 45 days after the patient has agreed to participate
  Evaluation of the prevalence of each mutation identified in the drainage vein of AVMs, with calculation of the exact 95% confidence interval.

SECONDARY OUTCOMES:
Evaluation of the imaging characteristics of cAVMs for each of the mutations identified. | Embolisation procedure (D0), i.e. a maximum of 45 days after the patient has agreed to participate
  Imaging characterisation of cAVMs for each of the mutations identified
Evaluate genetic mutations identified by liquid biopsies on the peripheral vein of AVMs. | Embolisation procedure (D0), i.e. a maximum of 45 days after the patient has agreed to participate
  determination of each mutation identified in the peripheral vein of AVMs
Assessment of the prevalence of each mutation identified by liquid biopsies on the peripheral vein of AVMs | Embolisation procedure (D0), i.e. a maximum of 45 days after the patient has agreed to participate
  Evaluation of the prevalence of each mutation identified in the peripheral vein of AVMs, with calculation of the exact 95% confidence interval.

CONTACTS AND LOCATIONS:
Locations (3):
- France (3):
  - University Hospital of Caen, Caen
  - Hôpital la Pitié-Salpêtrière, Paris
  - University Hospital of Rouen, Rouen

IPD SHARING:
Plan to Share IPD: No
The data provided will be the property of the sponsor and will be used solely for its own research activities.